CLINICAL TRIAL: NCT03129659
Title: Coronary CT Angiography for Improved Assessment of Suspected Acute Coronary Syndrome With Inconclusive Diagnostic Work-up
Brief Title: Coronary CT Angiography for Improved Assessment of Suspected Acute Coronary Syndrome
Acronym: COURSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Admir Dedic, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COURSE-11
Record Dates: First submitted 2017-04-16; First posted 2017-04-26 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Acute Coronary Syndrome; Chest Pain
Keywords: Coronary CT Angiography; High-sensitivity Troponin; Diagnosis
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT-group (Experimental): Coronary CT angiography
  Interventions: Diagnostic Test: Coronary CT Angiography

INTERVENTIONS:
Diagnostic Test: Coronary CT Angiography — Coronary CT angiography

SUMMARY:
Current evaluation of patients suspected of non-ST-elevation acute coronary syndrome is greatly dictated by the results of high-sensitivity troponins. In a substantial number of patients this approach does not provide a conclusive work-up. Patients typically present with slightly elevated high-sensitivity troponins without significant changes during serial sampling and no other clinical clues that can aid in determining the etiology of their chest pain complaints. Uncertainty remains about the optimal diagnostic management of these patients and they are often admitted to undergo invasive angiography. Coronary CT angiography can improve efficiency of clinical care in these patients by reducing unnecessary hospital admissions and invasive angiography. In this study, the investigators will investigate whether a diagnostic strategy comprising of early coronary CT angiography is more clinically efficient than standard optimal care in patients with an inconclusive work-up for non-ST-elevation acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency department with symptoms suggestive of NSTE-ACS. They do not fulfil criteria for either "rule-in" or "rule-out" NSTE-ACS based on serial sampling of high-sensitivity troponins and standard clinical work-up.

Exclusion Criteria:

* Inability or unwillingness to provide informed consent.
* History of proven CAD, defined as documented prior myocardial infarction, percutaneous coronary intervention or coronary artery bypass graft surgery.
* Previous examination with either invasive angiography or CCTA in the last 3 years.
* Clinical instability: clinical heart failure, hemodynamic instability, severe chest pain.
* CCTA-specific contra-indications:

  * Allergy to iodine contrast media
  * Pregnancy
  * Impaired renal function: estimated glomerular filtering rate <60% of the age-corrected normal values
  * Severe arrhythmia likely to affect image interpretation
  * BMI > 40
  * Inability to cooperate during the examination.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of coronary CT angiography to identify patients with NSTE-ACS. | 30 day
  Sensitivity and specificity of coronary CT angiography for the diagnosis of NSTE-ACS.

SECONDARY OUTCOMES:
Potential improvement of diagnostic accuracy with FFR-CT. | 30 day
  Off-line calculation of FFR-CT will be performed and the diagnostic accuracy for NSTE-ACS will be determined and compared to conventional coronary CT angiography.
Clinical characteristics of no obstructive coronary artery disease on CT. | 30 day
  To determine which clinical characteristics are predictive of not having obstructive coronary artery disease on CT.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amphia ziekenhuis, Breda, North Brabant
  - Erasmus MC, Rotterdam, South Holland

REFERENCES:
- [Derived] Arslan M, Schaap J, van Gorsel B, Aubanell A, Budde RPJ, Hirsch A, Smulders MW, Mihl C, Damman P, Sliwicka O, Habets J, Dubois EA, Dedic A. Coronary computed tomography angiography improves assessment of patients with acute chest pain and inconclusively elevated high-sensitivity troponins. Eur Radiol. 2025 Feb;35(2):789-797. doi: 10.1007/s00330-024-10930-1. Epub 2024 Aug 16. PMID 39150488
- [Derived] Arslan M, Schaap J, Van Gorsel B, Budde RP, Bekkers SC, Van Cauteren YJ, Damman P, Habets J, Dubois EA, Dedic A. Coronary CT angiography for improved assessment of patients with acute chest pain and low-range positive high-sensitivity troponins: study protocol for a prospective, observational, multicentre study (COURSE trial). BMJ Open. 2021 Oct 18;11(10):e049349. doi: 10.1136/bmjopen-2021-049349. PMID 34663657